CLINICAL TRIAL: NCT03477539
Title: Phase II Trial of Daratumumab for Transplant-Eligible Multiple Myeloma Patients
Brief Title: Daratumumab in Treating Transplant-Eligible Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1785; NCI-2018-00332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1785 (Other: Mayo Clinic in Florida); 17-004126 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-03-02; First posted 2018-03-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation; daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (daratumumab, ASCT, lenalidomide) (Experimental): CONSOLIDATION I: Patients receive daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2, and on days 1 and 15 of cycles 3-4. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION II: Beginning 8 weeks after completion of daratumumab cycle 2 or 4, patients undergo ASCT.
  MAINTENANCE: Within 14 days after completion of day 100 visit post-SCT, patients receive daratumumab IV on day 1 and lenalidomide PO daily on days 1-21. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients who are still maintaining response continue to receive daratumumab IV every 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Daratumumab; Drug: Lenalidomide

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase II trial studies how well daratumumab works in treating transplant-eligible patients with multiple myeloma. Daratumumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the percentage of patients achieving minimal residual disease (MRD) negativity by multiparameter flow cytometry (MPF) after autologous stem cell transplant (SCT) (at day 100) using pre-SCT daratumumab consolidation.

SECONDARY OBJECTIVES:

I. To determine percentage of patients achieving MRD negativity by MPF after 1 year of daratumumab+lenalidomide-based maintenance therapy.

II. To determine progression-free survival (PFS) for peri-SCT treatment with daratumumab.

III. To determine percentage of MRD negativity by MPF after pre-SCT consolidation with daratumumab.

IV. To determine safety profile of peri-SCT daratumumab with lenalidomide. V. To determine the overall response rate (ORR) of patients receiving peri-SCT daratumumab for MM.

VI. To determine the overall survival (OS) for patients receiving peri-SCT daratumumab for MM.

OUTLINE:

CONSOLIDATION I: Patients receive daratumumab intravenously (IV) on days 1, 8, 15, and 22 of cycles 1-2, and on days 1 and 15 of cycles 3-4. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION II: Beginning 8 weeks after completion of daratumumab cycle 2 or 4, patients undergo autologous stem cell transplant (ASCT).

MAINTENANCE: Within 14 days after completion of day 100 visit post-SCT, patients receive daratumumab IV on day 1 and lenalidomide orally (PO) daily on days 1-21. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients who are still maintaining response continue to receive daratumumab IV every 3 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Considered transplant eligible
* Pathologically confirmed diagnosis of multiple myeloma who are transplant eligible and have received any prior induction therapy (with or without maintenance)
* Measurable MRD in bone marrow within 28 days prior to registration (MPF method)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2 at registration
* Absolute neutrophil count (ANC) >= 1,000 cell/mm^3 without growth factor support, obtained =< 14 days prior to registration
* Platelets >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis < 50% or >= 30,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50%, obtained =< 14 days prior to registration
* Calculated or measured creatinine clearance >= 30 ml/min, obtained =< 14 days prior to registration
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome, in which case the direct bilirubin must be =< 1.5 X ULN, obtained =< 14 days prior to registration
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) =< 3 x ULN, obtained =< 14 days prior to registration
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 X ULN, obtained =< 14 days prior to registration
* Negative urine or serum pregnancy test for women of childbearing potential

  * NOTE: females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Provide informed written consent
* Measurable disease of multiple myeloma at the time specified by one of the following:

  * If no relapse prior to transplant, values obtained at the time of diagnosis
  * If disease relapse prior to transplant and the patient did not have treatment for the relapsed disease prior to transplant, the values obtained at the time of relapse immediately prior to the transplant.
  * If disease relapse prior to transplant and the patient did have treatment for the relapsed disease prior to transplant, the values obtained prior to this therapy, i.e., the time of relapse

Exclusion Criteria:

* Any previous ASCT for multiple myeloma (MM) (NOTE: Patient may have had prior stem cell collection before registration on the study)
* Any prior therapy with daratumumab
* Non-secretory MM or known amyloid light-chain (AL) amyloidosis
* Clinically significant active infection requiring intravenous antibiotics (=< 14 days prior to registration)
* >= grade 3 neuropathy and/or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Other prior malignancy

  * Exceptions:

    * Adequately treated basal cell or squamous cell skin cancer
    * Any in situ cancer
    * Adequately treated stage I or II cancer from which the patient is currently in complete remission, or
    * Any other cancer from which the patient has been disease free for at least 3 years
* Concurrent therapy considered investigational

  * NOTE: patients must not be planning to receive any radiation therapy (except localized radiation for palliative care that must be completed prior to starting cycle 1, day 1)
* Pregnant women
* Nursing women (lactating females are eligible provided that they agree not to breast feed while taking lenalidomide)
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Major surgery =< 4 weeks prior to registration
* History of stroke/intracranial hemorrhage =< 6 months prior to registration
* Clinically significant cardiac illness including New York Heart Association (NYHA) class III or class IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or >= grade 3 cardiac arrhythmias noted =< 14 days prior to registration
* Known human immunodeficiency virus positive (HIV+) patients
* Known hepatitis B or hepatitis C infection
* Exhibiting clinical signs of meningeal involvement of multiple myeloma
* Known severe chronic obstructive pulmonary disease or asthma defined as forced expiratory volume (FEV1) in 1 second less than < 60% of expected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Rate of minimal residual disease (MRD) negative response after autologous stem cell transplantation (ASCT) | At day 100 post ASCT
  MRD negative response after ASCT is defined as achievement of MRD negative status in the bone marrow by flow cytometry (multiparameter flow cytometry [MPF]) at the day 100 post ASCT visit. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. 95 percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
The rate of MRD negative response after pre-stem cell transplant (SCT) consolidation with daratumumab | Up to 3 years
  This will be estimated by the number of patients who achieve MRD negative status by flow cytometry (MPF) in the bone marrow after pre-SCT consolidation with daratumumab divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true rate of MRD negative response after pre-SCT consolidation with daratumumab will be calculated.
Rate of MRD negative response after 1 year (12 courses) of daratumumab and lenalidomide maintenance | At 1 year (12 cycles) of daratumumab and lenalidomide maintenance
  This will be estimated by the number of patients who achieve MRD negative status by flow cytometry (MPF) in the bone marrow after 1 year of maintenance therapy divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true rate of MRD negative response after 1 year of maintenance will be calculated.
Progression-free survival | From registration up to 3 years
  The distribution of progression-free survival will be estimated using the Kaplan-Meier method.
Survival time | From registration up to 3 years
  The distribution of survival time will be estimated using the Kaplan-Meier method.
Overall response rate | At day 100 post ASCT
  This will be estimated by the number of patients with an objective status of stringent complete responses, complete response, very good partial response, or partial response at the day 100 post ASCT assessment divided by the total number of evaluable patients. Response assessment will be in comparison to values obtained at the disease assessment at the time registration. Exact binomial 95% confidence intervals for the true overall response rate at day 100 post ASCT will be calculated.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
MRD assessment in blood and bone marrow | Up to cycle 18/16 months of treatment
  MRD assessment will be correlated between blood and bone marrow. Patients will be categorized as positive versus (vs.) negative MRD. The number of patients who have agreement between the 2 measures (both positive or both negative) will be assessed.
MRD assessed using flow cytometry (MPF) and next generation sequencing (NGS) | Up to cycle 18/16 months of treatment
  MRD assessment will be correlated between flow cytometry (MPF) and NGS. Patients will be categorized as positive vs. negative MRD for each measure. The number of patients who have agreement between the 2 measures (both positive or both negative) will be assessed.
Immune repertoire profiling | Up to cycle 18/16 months of treatment
  This will be assessed as continuous variables and their mutual change over time as assessed on the pre-specified time points will be correlated with response category to the treatment.
Antibody-dependent cellular phagocytosis and antibody-dependent cell-mediated cytotoxicity | Up to cycle 18/16 months of treatment
  These will be assessed as continuous variables and their mutual change over time as assessed on the pre-specified time points will be correlated with response category to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03477539/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03477539/ICF_002.pdf